CLINICAL TRIAL: NCT03255577
Title: Sentinel Lymph Node Biopsy After Neoadjuvant Chemotherapy in Patients Presenting With Locally Advanced Breast Cancer: A Prospective Study
Brief Title: Sentinel Lymph Node Biopsy After Neoadjuvant Chemotherapy For Locally Advanced Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-384
Record Dates: First submitted 2017-08-18; First posted 2017-08-21 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Locally Advanced Breast Cancer
Keywords: Sentinel Lymph Node Biopsy; 17-384
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Intervention Model Description: This will be a prospective single-arm study design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sentinel Lymph Node Biopsy (SLNB) (Experimental): The patients will undergo SLNB with dual tracer mapping using technetium-99m sulfur colloid and isosulfan blue dye, as is standard practice at our institution for cN1 patients. Than the SLNB procedure will be performed
  Interventions: Procedure: Sentinel Lymph Node Biopsy (SLNB)

INTERVENTIONS:
Procedure: Sentinel Lymph Node Biopsy (SLNB) — Sentinel Lymph Node Biopsy Patients with locally advanced breast cancer will undergo SLNB with dual tracer mapping followed by completion axillary lymph node dissection.

SUMMARY:
This study is being done to help the investigators determine how accurate the sentinel lymph node biopsy (SLNB) procedure is in identifying residual cancer cells after neoadjuvant chemotherapy in patients presenting with locally advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients over 18 years of age with biopsy-proven breast cancer
* Patients presenting with locally advanced disease in the breast (cT4) and/or in the nodes (cN2/N3) as assessed by clinical exam and imaging
* Patients presenting to surgery clinic after receipt of NAC at outside hospital with documentation of cT4 or cN2/3 disease on initial outside physical exam and imaging studies
* Patients receiving NAC and having a nodal complete clinical response as assessed by physical exam

Exclusion Criteria:

* Patients with a prior history of ipsilateral breast cancer
* Pregnant patients
* Patients with persistent palpable axillary nodes after NAC, as assessed by physical exam
* Patients not consenting to ALND

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 170 (Estimated)
Dates: Start 2017-08-17 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
The false negative rate of sentinel lymph node biopsy in patients with locally advanced breast cancer | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Barrio, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - BAPTIST ALLIANCE - MCI (Data Collection Only), Miami, Florida
  - Memorial Sloan Kettering at Basking Ridge (Consent and Follow Up), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only and Follow Up), Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent only and Follow Up), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm